CLINICAL TRIAL: NCT03470350
Title: MoTriColor: Phase I/II Study With Galunisertib (LY2157299) Combined With Capecitabine in Patients With Advanced Chemotherapy Resistant Colorectal Cancer and an Activated TGF-beta Signature
Brief Title: Galunisertib and Capecitabine in Advanced Resistant TGF-beta Activated Colorectal Cancer
Acronym: EORTC1615
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No study drug available. Same concept with new study drug will be explored in M19TGA study
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Vall d'Hebron Institute of Oncology (Other); Agendia (Industry); European Organisation for Research and Treatment of Cancer - EORTC (Network); Azienda Ospedaliera Niguarda Cà Granda (Other); Fundación para la Investigación del Hospital Clínico de Valencia (Other); University of Campania Luigi Vanvitelli (Other); University of Turin, Italy (Other); Eli Lilly and Company (Industry); Catalan Institute of Health (Other Government); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16TGA; 2016-002349-50 (EudraCT Number)
Record Dates: First submitted 2018-02-14; First posted 2018-03-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer Metastatic
Keywords: TGF-beta activatied
MeSH Terms: interventions — LY-2157299; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TGF-beta activated colorectal cancer (Experimental): TGF-beta activated advanced colorectal cancer treated with galunisertib and capecitabine
  Interventions: Drug: Galunisertib

INTERVENTIONS:
Drug: Galunisertib — treatment with capecitabine and galunisertib
  Other Names: Capecitabine

SUMMARY:
Part I of this study is designed to identify the recommended phase 2 dose (RP2D) of the combination regimen of galunisertib/capecitabine as second line treatment in patients with 5-FU or capecitabine resistant CRC. Part II is designed to obtain proof of principle of the galunisertib plus capecitabine combination in patients with chemo-resistant CRC. The combination of galunisertib plus capecitabine will be given as second line therapy in the phase II part of this study.

Patients with chemotherapy resistant activated TGF-β signature-like tumors will have received a fluoropyrimidine (5FU or capecitabine) in the first line of chemotherapy, usually combined with oxaliplatin and, depending upon local hospital preferences or national guidelines, also bevacizumab, or cetuximab/panitumumab if the tumor is KRAS wild type. Addition of galunisertib to capecitabine should thus result in reversal of unresponsiveness, which is the first step in exploring this concept in the clinic. Capecitabine can be used as single agent in advanced CRC and is thus attractive for this study concept. If proof of principle is achieved also other tumor types can be explored with this genetic makeup, such as non-small cell lung cancer (NSCLC) in second line of treatment after platinum doublet therapy in first line, usually cisplatin/carboplatin-pemetrexed in non-squamous and cisplatin/carboplatin-gemcitabine or cisplatin/carboplatin-paclitaxel in squamous type NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of CRC;
2. Disease progression or relapse upon first line of treatment (maximum lines of treatment is one for phase I and phase II of this study) for advanced CRC with fluoropyrimidine containing chemotherapy as single agent or in combination (combinations with oxaliplatin, irinotecan, bevacizumab and cetuximab/panitumumab are allowed);
3. Written documentation of activated TGF-β signature-like gene signature, as determined by the validated assay of Agendia;
4. Age ≥ 18 years;
5. Able and willing to give written informed consent;
6. WHO performance status of ≤ 1;
7. LVEF ≥ 55%;
8. Able and willing to undergo blood sampling for PK and PD analysis;
9. Able and willing to undergo tumor biopsies before start, during treatment and at the end of treatment
10. Life expectancy ≥ 3 months allowing adequate follow up of toxicity evaluation and anti-tumor activity;
11. Evaluable disease according to RECIST 1.1 criteria (measurable disease for the phase II part; evaluable disease is sufficient for the phase I part);
12. Minimal acceptable safety laboratory values

    1. ANC of ≥ 1.5 x 109 /L
    2. Platelet count of ≥ 100 x 109 /L
    3. Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALAT and ASAT ≤ 3.0 x ULN, or ALAT and ASAT ≤ 5 x ULN in patients with liver metastases
    4. Renal function as defined by serum creatinine ≤1.5 x ULN
    5. Creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula or MDRD);
13. Negative pregnancy test (urine or serum) for female patients with childbearing potential.

Exclusion Criteria:

1. Any treatment with investigational drugs within 30 days prior to receiving the first dose of investigational treatment;
2. Known or suspected dihydropirimidine dehydrogenase deficit (Mutant for DPD*2A genotype, 1236 GA genotype, 1679TG genotype and 2846A>T genotype);
3. Symptomatic or untreated leptomeningeal disease;
4. Symptomatic brain metastasis. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid therapy are allowed to enrol. Brain metastasis must be stable with verification by imaging (e.g. brain MRI or CT (<21 days before start of treatment) completed at screening demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive enzyme inducing anti-epileptic drugs or corticosteroids;
5. History of cardiac disease, including myocardial infarction within 6 months before study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension, major cardiac abnormalities, a predisposition for developing aneurysms including family history of aneurysms, Marfan syndrome, bicuspid aortic valve, or evidence of damage to the large vessels of the heart.
6. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral galunisertib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection);
7. Woman who are pregnant or breast feeding;
8. Unreliable contraceptive methods. Both men and women enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms);
9. Radio- or chemotherapy within the last 2 weeks prior to receiving the first dose of investigational treatment. Palliative radiation (1x 8Gy) is allowed;
10. Patients who have undergone any major surgery within the last 2 weeks prior to starting study drug or who would not have fully recovered from previous surgery;
11. Active infection requiring systemic antibiotics or uncontrolled infectious disease;
12. Patients with a known history of hepatitis B or C or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
13. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study;
14. Known hypersensitivity to one of the study drugs or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-24 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: The recommended phase 2 dose (RP2D) of galunisertib plus capecitabine in patients with chemotherapy resistant activated TGF-β signature-like CRC. | 6 months
Phase II: Response rate (RR) of galunisertib in combination with capecitabine in patients with chemotherapy resistant activated TGF-β signature-like CRC. | 15 months

SECONDARY OUTCOMES:
The incidence and severity of adverse events | 15 months
duration of response | 15 months
time to response | 15 months
overall survival (phase II only) | 15 months
progression free survival (phase II only) | 15 months
Plasma concentrations of galunisertib in combination with chemotherapy | 15 months
Gene alterations/expression profiles (e.g. baseline, relapse) in tumor tissue upon progression | 15 months
Baseline molecular status of potential predictive markers of tumor response | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: J Tabernero, Prof, Principal Investigator — VHIO; R Salazar, MD, PhD, Principal Investigator — ICO; R Bernards, Prof, Principal Investigator — Agendia; S Siena, Prof, Principal Investigator — ONCG; A Cervantes, Prof, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA; F Ciardiello, Prof, Principal Investigator — Unina2; A Bardelli, Prof, Principal Investigator — UNITO; S Tejpar, Prof, Principal Investigator — UZ Leuven
Locations (1):
- Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.motricolor.eu